CLINICAL TRIAL: NCT03727568
Title: Prospective, Randomised Study Comparing Two Different Methods of Transbronchial Cryobiopsy in the Interstitial Lung Diseases
Brief Title: Study Comparing Two Different Methods of Cryobiopsy in the Interstitial Lung Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: Marta Cuyás (Unknown)
Responsible Party: Principal Investigator, Kaid Darwiche, PD Dr. med Kaid Darwiche, Head Department of Interventional Pneumology, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RLK-Kryo-1; 18-7951-BO (Registry Identifier: Ethical Review Board University Clinic Essen)
Record Dates: First submitted 2018-10-22; First posted 2018-11-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryobiopsy: longer freezing time (Experimental): Group nº1: A total of 3 samples with a freezing time of 7 seconds at least for the first biopsy and a freezing time from ≥5 seconds for the following biopsies.
  Interventions: Procedure: Cryobiopsy
- Cryobiopsy: shorter freezing time (Experimental): Group nº 2: A total of 8 samples with a freezing time of 3 seconds at least for the first biopsy and a freezing time from <5 seconds for the following biopsies.
  Interventions: Procedure: Cryobiopsy

INTERVENTIONS:
Procedure: Cryobiopsy — In this study the investigators want to evaluate the diagnostic yield comparing 2 different techniques of performing cryobiopsy. A shorter freezing time and more number of biopsies vs a longer freezing time and less number of biopsies would be compared. Patients are randomised to the groups 1 or 2 immediate before the bronchoscopy.
  Group 1: a total of 3 samples with a freezing time of 7 seconds at least for the first biopsy and freezing time for 5 seconds or more for the followings biopsies Group 2: a total of 8 samples with a freezing time of 3 seconds at least for the first biopsy and freezing time for less than 5 seconds for the followings biopsies

SUMMARY:
Interstitial lung diseases (ILD) are a heterogeneous collection of more than 100 different pulmonary disorders. Surgical lung biopsie in combination with multidisciplinary discussion is recommend in combination to reach a consensus diagnosis when the initial clinical evaluation is inconclusive in the diagnosis of ILD. Cryobiopsy via bronchoscopy is approved for lung biopsies and allows harvesting of large tissue samples of excellent. This technique is not jet standardized. In this prospective randomised study the investigators want to evaluate the diagnostic yield comparing two different techniques of performing transbronchial cryobiopsy. In this study would be compared a shorter freezing time and more number of biopsies vs a longer freezing time and less number of biopsies.

DETAILED DESCRIPTION:
Design:

The investigators design a prospective randomised multicenter study to assess the diagnostic value of cryobiopsy in patients with suspected Idiopathic Interstitial Pneumonia by comparing two different interventional methods.

Patients with suspected ILD in which the clinical, radiological and BAL-data are insufficient to establish a definitive clinical diagnosis, requiring then tissue specimen to determine a diagnosis would be included.

Therefore this all patients will undergo transbronchial cryobiopsy. If a definitive diagnosis even after cryobiopsy and MDD cannot be made, SLB will be recommended.

For the cryobiopsies the 1.9 mm cryoprobe and ERBECRYO®2 with carbon dioxide will be used. All transbronchial cryobiopsies have to be obtained of one or two lobes of the same lung and in at least two different segments. The bronchopulmonary segment for the cryobiopsy will be selected based on the radiological features shown on a high resolution computed tomography (HRCT) of the chest. The areas with exclusively fibrotic changes should be avoided. After having touched the pleura with the cryopobe, the probe is retracted one to two centimetres and then in this position the freezing process will be initiated. The flexible bronchoscope with the inserted cryoprobe will be removed through the rigid bronchoscope after the sample was obtained.

The cryobiopsies can be performed in rigid or flexible bronchoscopy. The use of a Fogarty occlusion balloon is left to the discretion of the bronchoscopist.

Experimental Groups:

Group nº1: A total of 3 samples with a freezing time of 7 seconds at least for the first biopsy and a freezing time from ≥5 seconds for the following biopsies.

Group nº 2: A total of 8 samples with a freezing time of 3 seconds at least for the first biopsy and a freezing time from <5 seconds for the following biopsies.

Patient preselection:

Inclusion criteria

1. Inpatients with suspected ILD based on clinical and radiological features
2. Inpatients with probable pulmonary sarcoidosis without hilar or mediastinal lymph node enlargement
3. Male or female patients aged ≥18 years
4. Signed the informed consent

Exclusion criteria

1. Bleeding risk:

   1. Known predisposition to bleeding
   2. International randomised ratio (INR) >1,5,
   3. Elevated partial thromboplastin time (PTT)
   4. Platelet count < 80000/ul)
   5. Patients who required full-dose therapeutic anticoagulation or double antiplatelet therapy which can not be stopped as recommended before the cryobiopsy
2. Oxygen saturation < 90% with supported Oxygen 2l/min
3. Diffusing capacity (DLCO) <35% or FVC< 50%
4. Significant pulmonary emphysema
5. Severe cardiac disease (angina pectoris, acute myocardial infarction in the last 6 month, acute hearth failure)
6. Documented pulmonary hypertension PAP sys >50mmHg
7. Typical UIP-Pattern in HRCT

Patient's recruitment:

The recruited patients who present all characteristics of the inclusion criteria and none of the exclusion criteria and who signed the inform consent undergo cryobiopsy. All patients undergo a clinical evaluation.

After the clinical evaluation a MDD will take place. In the first MDD a provisional clinical diagnose is proposed. If a transbronchial cryobiopsy is indicated by the MDD, patients are randomised to the groups 1 or 2 immediate before the bronchoscopy.

Once the histological result is achieved, another MDD including the pathologist for establishing the definitive clinical diagnose take place. As all local pathologists of the participating centres are experienced in ILD, the samples are evaluated by the respective pathologist. If case of uncertainty, the samples can be evaluated by a second pathologist in one of the participating centres.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with suspected ILD based on clinical and radiological features
* Male or female patients aged ≥18 years
* Signed the informed consent
* Clinical indication to performed a lung biopsy in radiologically proven ILD

Exclusion Criteria:

* Bleeding risk:

  * Known predisposition to bleeding
  * International randomised ratio (INR) >1,5,
  * Elevated partial thromboplastin time (PTT)
  * Platelet count < 80000/ul
  * Patients who required full-dose therapeutic anticoagulation or clopidogrel or other thienopyridines
* Oxygen saturation < 90% with supported Oxygen 2l/min
* Severe bullous pulmonary emphysema
* Severe cardiac disease (angina pectoris, acute myocardial infarction in the last 6 month, acute hearth failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 2 years
  The investigator will assess the proportion of patients in which a definitive diagnosis is possible after Multi-Disciplinary Discussion

SECONDARY OUTCOMES:
Complications | 2 years
  Number of pneumothorax, bleeding and acute exacerbation.
Number of diagnostic samples | 2 years
Correlation between the suspected clinical diagnosis and the histological diagnosis | 2 years
Correlation between between radiological pattern and final diagnosis | 2 years
  The investigator want to evaluate the patient rate in which the radiological pattern could be confirmed by histological finding

CONTACTS AND LOCATIONS:
Overall Officials: Kaid Darwiche, Principal Investigator — Head of department of inteventionel pneumology, Ruhrlandklinik Essen
Locations (1):
- Ruhrlandklinik, Essen, North Rhine-Westphalia, Germany